CLINICAL TRIAL: NCT06895928
Title: A Phase II, Multicenter, Open-Label Study of Safety, Tolerability and Efficacy of SHR-A2102 for Injection in Combination With Other Antitumor Therapies in Patients With Advanced Solid Tumors
Brief Title: A Trial of SHR-A2102 With Other Antitumor Therapies in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-209
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Bevacizumab; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: SHR-A2102; Drug: Bevacizumab Injection; Drug: Adebelimab Injection; Drug: Ametinib Mesylate Tablets; Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: SHR-A2102 — SHR-A2102 for injection.
Drug: Bevacizumab Injection — Bevacizumab injection.
Drug: Adebelimab Injection — Adebelimab injection.
Drug: Ametinib Mesylate Tablets — Ametinib mesylate tablets.
Drug: Osimertinib Mesylate Tablets — Osimertinib mesylate tablets.

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A2102 with other antitumor therapies in advanced solid tumors to explore the reasonable dosage, safety and efficacy of SHR-A2102 for advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The age of signing the informed consent is 18 -70 years, regardless of gender.
2. At least one measurable lesion according to RECIST v1.1 criteria.
3. The ECOG score is 0 or 1.
4. Expected survival ≥12 weeks.
5. Good level of organ function.
6. Have the ability to give informed consent and to comply with the treatment plan.
7. Male subjects whose partners are women of childbearing age and female subjects who are fertile are required to use highly effective contraceptive methods.

Exclusion Criteria:

1. Inadequately treated central nervous system metastases or the presence of uncontrolled or symptomatic active central nervous system metastases.
2. Spinal cord compression not cured by surgery and/or radiotherapy.
3. Subjects with uncontrolled tumor-related pain.
4. Received antitumor therapy within 4 weeks before the start of the study.
5. Subjects with severe cardiovascular and cerebrovascular disease.
6. History of immunodeficiency, including a positive HIV test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From day 1 to 90 days after the last dose.
Serious adverse events (SAEs) | From day 1 to 90 days after the last dose.
Objective response rate (ORR) | About 2 years.

SECONDARY OUTCOMES:
Disease control rate (DCR) | About 2 years.
Duration of response (DOR) | About 2 years.
Progression free survival (PFS) | About 2 years.
Overall survival (OS) | About 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Cancer hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided